CLINICAL TRIAL: NCT06051279
Title: Pattern of Congenital Hypothyroidism in Newborns in Sidi-Galal Clinic Assiut Governorate.
Brief Title: Pattern of Congenital Hypothyroidism in Newborns.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma El Zahra Fathy Mohamed Abdelhady, resident physician at family medicine department, Assiut University
Other Study IDs: Pattern of CH
Record Dates: First submitted 2023-09-12; First posted 2023-09-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pattern of CH

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases with TNH: Newborns with raised TSH level and normal FT4 (the confirmed raised TSH cases after thyroid hormone screening) that return normal without intervention within one month after birth.
- Cases with permanent congenital hypothyroidism: Newborns with raised TSH level and low FT4 (confirmed cases after thyroid hormone screening)
- Control group: Control group with matched age and gender with normal TSH at birth according to the neonatal TSH screening. Matched normal neonates will be selected to be compared with transient neonatal hyperthrotropinemia cases and permanent congenital hypothyroidism cases for studying of the predictors of transient neonatal hyperthyrotopinemia.

SUMMARY:
1. Study the pattern of congenital hypothyroidism in newborns after positive newborn screening results.
2. Assess the characteristics of the cases (permanent congenital hypothyroidism and transient neonatal hyperthyrotopinemia).

DETAILED DESCRIPTION:
Thyroid hormone is essential for normal somatic growth and neurological development in infants and children. Deficiency of thyroid hormone in the first 2 years of life results in congenital hypothyroidism (CH). CH manifests by mental retardation and growth retardation in newborn.

Newborn screening (NS) for CH aims to early diagnosis and treatment of hypothyroidism. CH occurs about one in 3000-4000 infants . CH is suspected in neonatal screening when capillary thyroid-stimulating hormone (TSH) concentrations are elevated (>15 mU/L in Germany). The diagnosis is confirmed by measuring venous TSH and free thyroxine levels (FT4) concentrations before the start of treatment.

CH can be classified into permanent or transient congenital hypothyroidism (TCH). While CH is a persistent deficiency of thyroid hormones that requires lifelong treatment, TCH is a temporary deficiency that reverts to normal concentrations with proper medical management, usually during the first few months of life and not after the age of 3 years.

Transient neonatal hyperthyrotropinemia (TNH) is defined as temporary postnatal elevation of TSH levels (10 mIU/L-20 mIU/L) with normal FT4 levels but TSH returning to normal (<10 mIU/L) when measured at 14 d of life. It is important to recognize TNH as these newborns have a higher risk of developing permanent hypothyroidism with repercussion on developmental status. Thus, we aimed at evaluating the neonatal and maternal factors associated with TNH . So that, identifying these factors may be considered as an appropriate strategy to prevent these possible disorders. There is a gap in studying the prevalence and the predictors of transient neonatal hyperthyrotropinemia particularly in Assiut Governorate.

ELIGIBILITY:
Inclusion Criteria:

* For the case series study: all positive newborns cases with raised TSH level (the confirmed raised TSH cases after thyroid hormone screening) within one month after birth will be taken during one year.
* For the secondary outcome to study the predictors of permanent congenital hypothyroidism and transient neonatal hyperthyrotropinemia, control group with matched age and gender with normal TSH at birth according to the neonatal TSH screening will be taken. Matched normal neonates will be selected to be compared with permanent congenital hypothyroidism cases and transient neonatal hyperthrotropinemia cases.

Exclusion Criteria:

* Cases that refused to participate in research.
* Cases that missed for follow up.

Ages: 15 Days to 2 Months | Sex: All
Age Groups: Child
Study Population: Cases: Newborn with TSH (the confirmed raised TSH cases after thyroid hormone screening) within one month after birth, both transient neonatal hyperthyrotropinemia cases and permanent congenital hypothyroidism included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Pattern of congenital hypothyroidism in newborns after positive newborn screening results. | through study completion, an average of 1 year
  The data will be collected from the records of laboratory investigation to assess the pattern of congenital hypothyroidism

SECONDARY OUTCOMES:
Predictors of permanent congenital hypothyroidism and transient neonatal hyperthyrotropinemia as neonatal, obstateric and maternal factors. | through study completion, an average of 1 year
  Determine if studied neonates on breastfeeding or not and have sufficient feeding signs or not by asking the child caregiver
Characteristics of studied newborns in all types of congenital hypothyroidism in Sidi-Galal clinic as in feeding, nutritional status and growth parameters. | through study completion, an average of 1 year
  Determine if studied neonates on breastfeeding or not and have sufficient feeding signs or not by asking the child caregiver